CLINICAL TRIAL: NCT03883009
Title: Understanding the Drivers of Surgical Site Infection: Investigating and Modeling the Swissnoso Surveillance Data
Acronym: WATUSSI
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Patient Safety Foundation (Unknown); Lucerne University of Applied Sciences and Arts (Unknown); University of Bern (Other); Swissnoso National Center for Infection Control (Unknown); Central Institute of Valais Hospitals (Unknown); University Hospital, Basel, Switzerland (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 32003B_179500
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Surgical Site Infection
Keywords: Epidemiology; Modeling; Risk factors; Surgical site infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical site infection (SSI) is the most common healthcare-associated infection, multifactorial in nature, and a typical preventable harm. Many healthcare systems require hospitals to determine the corresponding infection rates as a quality indicator and often stipulate public reporting of these data. Several agencies, among them the World Health Organization (WHO) and the U.S. Centers for Disease Control and Prevention (CDC), have issued evidence-based prevention guidelines. Despite efforts in implementing best practice, SSI continue to be a relevant complication of modern surgical procedures and generate enormous costs for the healthcare system. Moreover, prevention guidelines acknowledge that the evidence backing their recommendations is low to moderate in most cases, which is partly due to the complexity of SSI pathogenesis.

Swissnoso, the Swiss expert group for infection prevention and hospital epidemiology, oversees the nationwide collection of data on select procedures and the associated SSI. Since the inception of this dedicated surveillance in 2009, more than 300'000 procedures have been included and the corresponding patients were followed to ascertain SSIs. Although primarily conceived as a national surveillance system and then used for public reporting starting in 2014, Swissnoso is a prime data source for better understanding the epidemiology of SSI.

Here, the investigators seek to raise the quality of evidence behind future prevention guidelines. For this purpose, the investigators will move from a risk factor analysis for SSI (of which a substantial part occurs after patient discharge from the hospital, rendering surveillance difficult) to the collection of additional data (in order to better characterize certain determinants of SSI and their recognition) and, finally, to a mathematical model (which will simulate the probability of developing SSI so the investigators can test what may modulate this risk).

DETAILED DESCRIPTION:
Aim 1: Descriptive epidemiology and risk factors for (post-discharge) SSI: using the Swissnoso SSI Surveillance data, the investigators will determine patient and institution level risk factors for SSI in Switzerland (with a focus on those occurring post-discharge), explore protective factors (such as antimicrobial prophylaxis and its timing), and describe the epidemiology of SSI in terms of time of occurrence, microbiology, severity, patient outcome, and variation by procedure type, case-mix, and hospital size.

Aim 2: Determinants of SSI: The investigators will investigate determinants of SSI in the following three areas:

A) The surveillance system itself and how the thoroughness of the surveillance process correlates with reported SSI rates; B) The operating room ventilation system and how its parameters correlate with SSI rates; and C) A healthcare institution's perceived culture of safety and how it correlates with infection rates.

To do so, the investigators will enhance and complement the Swissnoso data with new information at the institution level.

Aim 3: A mathematical model of surgical site infection: the investigators will construct a mathematical model that simulates SSI pathogenesis based on data from Swissnoso and other sources, and assesses the impact of different preventive measures. Interventions will be ranked according to the simulated reduction of SSI rates in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* All cases included in the Swissnoso SSI Surveillance system are eligible for the analyses.

Exclusion Criteria:

* If a patient opts to withdraw consent to participating in the Swissnoso SSI Surveillance, his/her data is removed from the surveillance dataset.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Swissnoso SSI Surveillance: Nationwide surveillance system with 172 participating hospitals collecting data on patients who undergo select surgeries as defined by Swissnoso. Since 2009, information on 318'000 surgical procedures has been captured (database extract February 2017).
Sampling Method: Non-Probability Sample
Enrollment: 318000 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Surgical site infection rate | During 30 days after surgery (or 12 months after surgery with implants)
  Number of surgical site infection per number of corresponding surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Marschall, Prof.Dr.med., Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland